CLINICAL TRIAL: NCT04454281
Title: Topical Naloxone Hydrochloride as a Diagnostic Tool for Ocular Neuropathic Pain
Brief Title: Topical Naloxone to Diagnose Ocular Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seema Capoor (Other)
Responsible Party: Sponsor-Investigator, Seema Capoor, Principal Investigator, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 48303
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Dry Eye Syndromes; Neuropathic Pain
MeSH Terms: conditions — Dry Eye Syndromes; Neuralgia | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Naloxone HCl Low dose: 0.02 mg (Experimental): This arm will receive 0.02 mg naloxone hcl on the experimental visit and balance salt solution on the control visit.
  Interventions: Drug: Naloxone Hydrochloride 0.4 MG/ML
- Naloxone HCl High dose: 0.08 mg (Experimental): This arm will receive 0.08 mg naloxone hcl on the experimental visit and balance salt solution on the control visit.
  Interventions: Drug: Naloxone Hydrochloride 0.4 MG/ML

INTERVENTIONS:
Drug: Naloxone Hydrochloride 0.4 MG/ML — Drug will be topically applied to the corneal surface then study evaluations will ensue.

SUMMARY:
Chronic ocular neuropathic pain may be misdiagnosed as dry eye disease. Our study aims to identify a population with previous monocular trauma and dry eye symptoms and differentiate neuropathic from dry eye pain using topical corneal naloxone hydrochloride.

DETAILED DESCRIPTION:
Dry eye is a ubiquitous and debilitating ocular condition that affects tens of millions in the United States (DEWS, 2007). However, there is increasing evidence that the symptoms of dry eye overlap with the distinct condition of ocular neuropathic pain, and that many patients given a dry eye diagnosis are mislabeled (Galor, 2017). These shared symptoms include but are not limited to: hypoesthesia, hyperalgesia, and allodynia. According to the 2017 DEWS II (Dry Eye Workshop) pain and sensation report by the Tear Film and Ocular Surface Society, neuropathic pain can manifest itself in the eye and may present similarly to dry eye, but should not be classified as such (Belmonte, 2017). Our study aims to further characterize this distinction by translating the rodent model of latent sensitization to the human eye.

Latent sensitization is a model of chronic pain that reproduces both its episodic nature and its sensitivity to stress. It can be induced by an array of insults and follows a characteristic time course in which a hyperalgesic pain phase is followed by pain remission phase. Of clinical relevance, administration of mu-opioid antagonists (i.e. naloxone) during the remission phase reinstates animal pain behavior and physiologic reflexes to peak levels seen in the hyperalgesia phase (Marvizon, 2015). This phenomenon suggests that the animals are in a state of latent sensitization that can be unmasked by blocking the activity of the opioid signaling pathway through compounds like naloxone hydrochloride. Furthermore, the undulating course of chronic pain syndromes can be mimicked by introducing environmental and physical stressors that trigger and exacerbate pain states (Marvizon, 2015).

Neuropathic pain is a common cause of chronic pain. It is defined by the International Association for the Study of Pain as pain that arises as a direct consequence of a lesion or disease affecting the somatosensory system. In contrast, nociceptive pain is produced by the normal function of nociceptors. Hence, neuropathic lesions do not necessarily involve the nociceptive pathway; instead, they can involve other somatosensory pathways including tactile, mechanical, and thermal pathways. These lesions manifest allodynia-a central pain sensation following a normally non-painful stimuli and a clinical hallmark of neuropathic pain. In the eye, allodynia may manifest as non-specific dry-eye-like-symptoms to stimuli including wind, temperature change, and humidity (Galor, 2017).

Hyperalgesia is a heightened pain sensation to a normally painful stimulus and is another hallmark of neuropathic pain. Importantly, hyperalgesia is a symptom of both neuropathic and nociceptive pain, however the pathophysiologies are distinct. Neuropathic hyperalgesia is a sustained phenomenon that arises from neuronal remodeling and sensitization of nociceptive peripheral and/or central nerves. In distinction, nociceptive hyperalgesia arises from inflammatory cytokine mediators that sensitize nociceptors and resolves after the conclusion of inflammation. Given all of this, it can be difficult to clinically differentiate the two forms of hyperalgesia; similarly, it can be difficult to differentiate between neuropathic and nociceptive pain.

In our murine model (Cho, 2019), we study latent sensitization of the eye after injuring the cornea with an alkali solution. We find that pain behavior (quantified by the number of eye wipes in thirty seconds after the topical administration of 2M NaCl to the corneal surface) peaks at day 10 post injury and returns to baseline by day 14 post injury (figure 3.1; next page). Topical administration of naloxone (100uM, one drop), reinstated peak pain behavior 16 weeks after initial corneal surface injury (figure 3.2; next page).

We hypothesize that our patient population with monocular trauma and dry eye symptoms mirrors our murine model. The monocular trauma represents the initial corneal surface injury, and the dry eye symptoms represent the breakthrough pain. It is important to note that in other models of latent sensitization, peak pain responses can be reinstated by stressors other than opioid antagonism. Specifically, novel environment stressors and forced swims reproduce peak pain behavior experienced in the hyperalgesic phase. In a similar way, our patient population endorses exacerbation of dry eye symptoms in the setting of stress, sleep, and environmental changes.

Our study aims to differentiate dry eye disease from ocular neuropathic pain by testing the latent sensitization model in the human eye. Given that there is good data to suggest chronic pain states, including our ocular model, can be masked by upregulation of the mu-opioid receptor signaling pathway, we hypothesize that our naloxone hydrochloride drop will induce a hyperalgesic response to hypertonic saline in a population with dry eye diagnosis and monocular trauma. We believe a topical naloxone ophthalmic drop is a potentially easy, cheap, and safe diagnostic tool for ocular neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* monocular trauma
* dry eye disease diagnosis

Exclusion Criteria:

* any pathology that might contribute to ocular pain, including corneal surface ulcers, uveitis, or other chronic inflammatory processes
* any current corneal surface pathology
* history of bilateral ocular trauma
* currently taking any of the following medications: TCAs, opioids, gabapentin, SNRIs
* pregnant nor breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Pain Response to Hypertonic Saline (Muro 128) drop | Immediately after hypertonic drop administered. Measured during both study visits, thus through study completion, an expected average of 4 weeks.
  The pain response is graded using a Visual Analog Scale (VAS) survey. It is graded 1-10; 10 indicates the most severe pain.

SECONDARY OUTCOMES:
Ocular Surface Disease Index | At any point during study visit. Measured during both study visits, thus through study completion, an expected average of 4 weeks.
  This 12 question survey measures your recent dry eye symptoms using the ocular surface index scale. The scale has a low score of 10 and high score of 100. A higher score means you have worse dry eye symptoms.
Slit Lamp Biomicroscopy | Before and after hypertonic saline drop. Measured during both study visits, thus through study completion, an expected average of 4 weeks.
  This test examines many areas of your eye (cornea, lids, inner eye) using a microscope.
Flourescein corneal examination | Before and after hypertonic saline drop. Measured during both study visits, thus through study completion, an expected average of 4 weeks.
  A yellow staining dye will be applied to your cornea that will allow us to examine the structural integrity of your cornea.
intraocular pressure | Before and after hypertonic saline drop. Measured during both study visits, thus through study completion, an expected average of 4 weeks.
  Intraocular pressure will be measured via Tono-Pen.
visual acuity | Before and after hypertonic saline drop. Measured during both study visits, thus through study completion, an expected average of 4 weeks.
  will be measured using ETDRS letter grading system. Your grade will depend on your ability to read small print.

CONTACTS AND LOCATIONS:
Overall Officials: Seema Capoor, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No